CLINICAL TRIAL: NCT05555043
Title: Comparison of Clinical Outcomes Between GentleWave® and Biolase®: A Randomized Controlled Trial
Brief Title: Comparison of Clinical Outcomes Between GentleWave® and Biolase®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-2960
Record Dates: First submitted 2022-09-19; First posted 2022-09-26 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Endodontic Disease; Periapical Diseases; Periapical Periodontitis; Root Canal Infection
MeSH Terms: conditions — Dental Pulp Diseases; Periapical Diseases; Periapical Periodontitis | interventions — Therapeutic Irrigation

STUDY DESIGN:
Intervention Model Description: In this block-randomized, single-blinded, randomized control trial, 120 participants will be recruited with 40 participants allocated to the GentleWave System treatment group, 40 participants allocated to the Waterlase treatment group, and 40 participants allocated to a control group receiving commonly used passive ultrasonic irrigation treatment.
Who Masked: Outcomes Assessor
Masking Description: This is a single blinded study. Following randomization, the participant and treating clinician will not be blinded from the treatment. Reviewers of all data collected will be blinded to the treatment modality provided.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Control group (Active Comparator): Participants receive passive ultrasonic irrigation for endodontic irrigation treatment and will be followed for 12 months after treatment to assess radiographic healing of the periapex and clinical healing of the tooth.
  Interventions: Device: Irrisafe ip
- GentleWave group (Experimental): Participants receive GentleWave System for endodontic irrigation treatment and will be followed for 12 months after treatment to assess radiographic healing of the periapex and clinical healing of the tooth.
  Interventions: Device: GentleWave System
- Waterlase group (Experimental): Participants receive Waterlase iPlus for endodontic irrigation treatment and will be followed for 12 months after treatment to assess radiographic healing of the periapex and clinical healing of the tooth.
  Interventions: Device: Waterlase iPlus

INTERVENTIONS:
Device: Irrisafe ip — This portion of endodontic treatment includes chemical disinfection of the root canal system with these different devices that activate the disinfection solution and distribute it throughout the root canal system with ultrasonic energy.
  Other Names: Passive ultrasonic irrigation
  Arms: Control group
Device: GentleWave System — Prepare, clean and irrigate root canals including activation of the disinfection solution and distribution throughout the root canal system.
  Other Names: Sonic cleaning and irrigation
  Arms: GentleWave group
Device: Waterlase iPlus — Prepare tooth and root canal, including enlargement, to debride, clean and disinfect after endodontic treatment.
  Other Names: Powered Laser Surgical Instrument
  Arms: Waterlase group

SUMMARY:
Introduction: In the US, 15 million root canal treatments (RCTs) are carried out annually. Success rates decrease with conventional chemo-mechanical root canal preparation techniques used on teeth with periapical radiolucencies associated with bacterial presence. New irrigation modalities, such as the GentleWave® System (GWS) and Waterlase iPlus® (WL), have been developed to overcome limitations and improve RCT success rates.

Hypotheses: (1) GWS and WL provide superior clinical outcomes compared to conventional RCT using passive ultrasonic activation (PUI). (2) GWS and WL are acceptable treatment modalities for clinicians and patients.

Aims: (1) Estimate probability of success of GWS, WL, and conventional RCT with PUI. (2) Evaluate clinician and patient experiences of the different techniques.

DETAILED DESCRIPTION:
This is a single-blinded, block randomized control trial study, 120 participants will be recruited with 40 participants randomly allocated to the GWS treatment group, 40 randomly allocated to the WL treatment group, and 40 randomly allocated to the control group (CG) receiving PUI treatment (Fig 1). Participants will be selected consecutively based on our inclusion and exclusion criteria. Participants will be recruited and treated at a single site, the University of North Carolina at Chapel Hill Adams School of Dentistry (UNC-CH ASoD) Endodontic Clinic.

There will be an initial baseline/screening appointment that may or may not develop into the first treatment appointment, followed by a potential second treatment appointment to complete treatment as per current treatment protocols in the Endodontic Clinic. Then participants will be followed for 12 months to evaluate clinical and radiographic healing of periapical lesions. Investigators will also assess clinician and patient opinion of the treatment modality employed in addition to calculation of a cost-time ratio.

Patients will receive endodontic treatment for endodontic infections with potential improvements in procedure outcomes, number of visits, and patient intraprocedural comfort. There are the same risks for any root canal procedure that can include intraprocedural or postoperative sensitivity, inflammation infection, numbness, intraprocedural or postoperative pain, reaction to materials used, sodium hypochlorite extrusion, instrument fracture, or perforation. The investigators will manage these risks through execution of proper instrument usage and adherence to clinical protocols.

The investigators do not anticipate difficulty in recruiting the required number of study participants based on the number of patients seen annually. Each week, approximately fifty patients are seen in the ASoD clinic for endodontic treatment, of which at least 50% meet the inclusion criteria for our study. There are nine trained residents in endodontics who carry out approximately five-six treatments per week. Nevertheless, all subjects are free to withdraw from participation at any time, for any reason, specified or unspecified, and without prejudice. A subject may leave at any time if the subject and/or investigator feel that it is not in the subject's best interest to continue.

Study participants will be consecutively recruited from the Endodontic Clinic at UNC-CH ASoD. Specifically, they will be patients seeking endodontic treatment at ASoD. At the consult/treatment appointment, screened potential participants meeting the inclusion/exclusion criteria will be informed of the study and potential treatment modalities by a member of the research team who is not the treating clinician. Patients will be given adequate time to decide if they would like to participate. Once a participant consents/assents to participation in the study, they will be randomly allocated to either the control group, GentleWave treatment group, or the Waterlase treatment group in a block randomized manner. Once a participant is assigned a treatment, the treatment will take place at the same appointment as the baseline/screening appointment or scheduled for another appointment. Treatment will be completed in one or possibly two appointments. Thereafter, the patient will be scheduled for a 12-month follow up visit to evaluate clinical and radiographic healing of the periapical lesion and tooth. This follow-up appointment, depending on the amount of treatment appointments required to complete treatment, may be the second, third, or fourth appointment.

Patients who agree to participate in the study will be randomized to either the GWS, WL, or control groups. As previously mentioned, each treatment group consists of 40 patients. Eight blocks of fifteen treatments (five of each treatment type) will be used. Once a patient consents/assents to participation in the study, a third party will be contacted who has access to the block randomization and they will inform the research team which treatment the patient is to undergo. This will help with organization of the treatment room with the appropriate equipment. Patient details and treatment allocation will be recorded on a password-protected Excel spreadsheet.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 14 years of age or older (maximum of 99 years of age)

  o Participants 14 years of age or older are expected to have permanent teeth erupted in full permanent dentition with close apices
* The subject tooth is indicated for root canal treatment

  * One tooth indicated per participant
  * Permanent tooth requiring root canal treatment which are deemed restorable
  * Teeth exhibiting pulpal pathosis (irreversible pulpitis, pulpal necrosis, previously initiated root canal treatment) and apical periodontitis (with radiographic demonstration of periapical bone loss)
* Patient-signed informed consent/assent form
* Patients display good compliance o Patient is determined cooperative by provider during initial exam and radiographic acquisition

Exclusion Criteria:

* Patients allergic to local or topical anesthetics, heart disease (pacemakers, implantable defibrillators), lung disease, bleeding disorders, immune system deficiency
* Subject tooth is not clinically restorable (prosthetically or periodontally)

  * Mobility scores greater than or equal to 2
  * Periodontal pocket depths greater than or equal to 6mm
  * Cracks with radicular extension, vertical root fracture or horizontal - oblique fracture
* Subject tooth with open or incomplete apices (apical diameter greater than 1mm)
* Subject tooth has insufficient tooth structure to create GWS platform
* Subject tooth has external cervical root resorption
* Subject tooth has signs of dens invaginatus
* Subject tooth has signs of a palatogingival groove
* Subject tooth has root(s) which communicate with the maxillary antrum
* Patient has nonodontogenic facial pain
* Patient requires multiple teeth to be endodontically treated

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Periapical index score | 12 months
  A combination of the clinical findings and Periapical Index Scores (PAI) score will be used to determine the primary outcome measure as healed, healing, or diseased as per the following descriptions:
  (i) Healed: Clinical normalcy other than tenderness to percussion accompanied by PAI scores of 1 or 2 (ii) Healing: Clinical normalcy other than tenderness to percussion accompanied by a reduction in the size of the periradicular lesion denoted by a reduction in the PAI score (iii) Diseased: The presence of clinical signs and symptoms accompanied by a PAI score of 3 or higher or an increase in the PAI score This is a scale of 1-5, where generally a higher number means poorer healing.

SECONDARY OUTCOMES:
Qualitative data from patient and provider questionnaires about treatment procedure | from time of treatment completion to 12-month follow-up appointment, assessed up to 12 months
  Secondary analyses will include summaries of questionnaires. Questionnaires will be sent out to participants after after treatment is completed with various structured questions utilizing the Likert scale. For example, questions will consist of "During my endodontic treatment, I felt comfortable (strongly disagree (1) to strongly agree (5)". Furthermore, for selected participants, semi-structured interview transcripts will undergo qualitative analysis which will consist of coding transcripts based on both deductive and inductive topics related to experiences with treatment. Data from the groups will be triangulated to assess convergence and possible differences in perceptions and preferences. Analysis will include examining co-occurrences of codes with a final report describing primary topics across all data. Specialized qualitative software, MAXQDA, will be used for coding, analysis, and generating final products such as matrices and diagrams.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Karunanayake, BDS, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Univeristy of North Carolina Adams School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.